CLINICAL TRIAL: NCT03879668
Title: Palli-MONITOR: A Phase II Mixed-Methods Study to Implement and Test the Electronic Version of the Integrated Palliative Care Outcome Scale (eIPOS) in an Specialist Palliative Home Care
Brief Title: Monitoring of Palliative Care Needs in Specialized Palliative Home Care Using the Electronic Version of the Integrated Palliative Care Outcome Scale
Acronym: Palli-MONITOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Claudia Bausewein, Professor for Palliative Medicine, Ludwig-Maximilians - University of Munich
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 01VSF17014
Record Dates: First submitted 2019-03-11; First posted 2019-03-19 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Advanced Disease
Keywords: Advanced disease; Specialised outpatient palliative care; IPOS; Electronical monitoring

STUDY DESIGN:
Intervention Model Description: Convergent mixed methods design: Quantitative quasi-experimental study with retrospective and prospective control group; Qualitative interviews with patients and focus groups with professionals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- eIPOS (Experimental): The cohort will include all participants who are cared for by the participating specialist palliative home care teams when implementing eIPOS.
  Interventions: Device: eIPOS
- Historic control (No Intervention): The cohort will include all participants that were cared for by the participating specialist palliative home care teams in the last 6 months before the implementation of eIPOS.
- Prospective control (No Intervention): The cohort will include participants who are in the care of the participating specialist palliative home care teams at the same time as the eIPOS group, but who do not use eIPOS.

INTERVENTIONS:
Device: eIPOS — Electronic version of IPOS
  Arms: eIPOS

SUMMARY:
In palliative care, the Integrated Palliative Care Outcome Scale (IPOS) is widely used as a patient reported outcome measure (PROM) and covers patients' main concerns, common symptoms, patient and family distress, existential wellbeing, sharing feelings with family, information received, and practical concerns. The IPOS is validated for patients with advanced cancer or non-cancer disease and is available as patients and professional carer version.

The implementation of a PROM in the home care setting is more challenging compared to the inpatient setting.

Palli-MONITOR will develop, implement and test the feasibility of an internet-based real-time monitoring of palliative needs of patients with advanced diseases using the electronic version of IPOS (eIPOS) including a clinical decision support tool for specialist palliative home care.

The project is conducted in two parts:

1. A pilot study to develop an electronical monitoring that is acceptable for both palliative patients and professionals of specialist palliative home care teams.
2. A feasibility study to implement and test eIPOS in specialist palliative home care teams.

DETAILED DESCRIPTION:
In palliative care, the Integrated Palliative Care Outcome Scale (IPOS) is widely used as a patient reported outcome measure. IPOS covers patients' main concerns, common symptoms, patient and family distress, existential wellbeing, sharing feelings with family, information received, and practical concerns. IPOS is validated for patients with advanced cancer or non-cancer disease and is available as patients and professional carer version.

The implementation of a PROM in the home care setting is more challenging compared to the inpatient setting. Furthermore, IPOS currently only exists as a paper version. If patients complete the IPOS at home, there is a potential delay until the home care team receives the information and a potential benefit through patient reported outcome measurement might be missed.

Palli-MONITOR will develop, implement and test the feasibility an internet-based real-time monitoring of palliative needs of patients with advanced disease using the electronic version of IPOS (eIPOS) including a clinical decision support tool for specialist palliative home care.

The project is conducted in two parts (phase I and phase II). Phase I will consist of two components and serve as a pilot study: a qualitative part and a cross-over randomised controlled trial (RCT). In the qualitative part, the investigators will conduct semi-structured interviews and focus groups with patients and professionals of the participating specialist palliative home care teams. In the RCT, the investigators will determine the validity of the eIPOS in comparison to IPOS in paper version. The investigators will also develop an evidence-based Clinical Decision Support Tool (CDS), using guidelines and a Delphi study for evaluation of the proposed CDS.

Phase II (study design described in more detail below) will serve as a feasibility study and consist of an observational case-control study as well as a qualitative part, which again will include semi-structured interviews and focus groups.

This mixed-methods approach will help to implement eIPOS while ensuring at the same time that the quality of palliative care during the process will meet at least the current standards.

ELIGIBILITY:
Inclusion Criteria:

* Participants cared for by one of the participating specialist palliative home care teams
* Participants who have the capacity to give informed consent to participate the study in writing and are able to participate in research
* Participants who are not too distressed or ill to participate in the study

Exclusion Criteria:

* Participants with cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Recruitment rates | 1 year
  The recruitment rates of each specialist palliative home care teams will be calculated as the percentage of eligible participants who agreed to participate in the study divided by the total number of eligible participants approached to participate in the study.
Acceptance of electronical monitoring | up to 4 weeks after enrollment
  Based on qualitative data
Technical feasibility of electronical monitoring: Integrated Palliative Care Outcome Scale | up to 4 weeks after enrollment
  Completeness of the electronic Integrated Palliative Care Outcome Scale (eIPOS). IPOS includes 10 symptoms and 7 questions on patients and carers emotional situation, spiritual concerns, and provision of information and support. Five answer options for each question are possible (scored 0 to 4; higher scores indicate higher burden). The overall IPOS score is the sum of the scores from each of the 17 questions. The overall IPOS score can therefore range from zero to 68.
Influence of electronical monitoring on provided care | up to 4 weeks after enrollment
  Assess care modifications consecutive of initial care

SECONDARY OUTCOMES:
Palliative needs (IPOS) | up to 4 weeks after enrollment
  Change in palliative care needs and specific symptoms assessed with the Integrated Palliative Care Outcome Scale (IPOS). IPOS includes 10 symptoms and 7 questions on patients and carers emotional situation, spiritual concerns, and provision of information and support. Five answer options for each question are possible (scored 0 to 4; higher scores indicate higher burden). The overall IPOS score is the sum of the scores from each of the 17 questions. The overall IPOS score can therefore range from zero to 68.
EORTC QLQ-C15-PAL | At baseline and 2 weeks
  Change from baseline in quality of life (at 2 weeks) assessed with the European Organization for Research and Treatment of Cancer (EORTC) questionnaire of life quality (QLQ). The adapted version for palliative (PAL) cancer care patients will be used.
  One item, scored from 1 to 7 (higher scores indicate better quality of life), gives an overall score corresponding to the quality of life that the patient feels he or she has.
Symptom burden (ESAS) | At baseline and 2 weeks
  Change from baseline in symptom burden (at 2 weeks) assessed with the Edmonton Symptom Assessment Scale (ESAS). ESAS includes 9 common symptoms. The severity of each symptom is rated from 0 to 10 on a numerical scale (higher scores indicate higher intensity).
Unplanned hospital submissions | up to 3 weeks after enrollment
  Number of patients with unplanned hospitalization, assessed from medical record

CONTACTS AND LOCATIONS:
Locations (1):
- Katerina Hriskova, München, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burner-Fritsch I, Kolmhuber S, Hodiamont F, Bausewein C, Hriskova K. Implementing ePROM in specialist palliative home care: the professionals' perspective - a mixed-methods study. Palliat Care Soc Pract. 2023 Aug 6;17:26323524231186827. doi: 10.1177/26323524231186827. eCollection 2023. PMID 37560175
- [Derived] Bolzani A, Kupf S, Hodiamont F, Burner-Fritsch I, Bausewein C, Ramsenthaler C. Measurement equivalence of the paper-based and electronic version of the Integrated Palliative care Outcome Scale (IPOS): A randomised crossover trial. Palliat Med. 2023 May;37(5):760-770. doi: 10.1177/02692163231157871. Epub 2023 Mar 1. PMID 36856258
- [Derived] Bolzani A, Ramsenthaler C, Hodiamont F, Burner-Fritsch IS, Bausewein C. Monitoring of Palliative Care Symptoms and Concerns in Specialized Palliative Home Care Using an Electronic Version of the Integrated Palliative care Outcome Scale (Palli-MONITOR): protocol for a mixed-methods study. BMJ Open. 2021 Jun 1;11(6):e042266. doi: 10.1136/bmjopen-2020-042266. PMID 34078632

DOCUMENTS (1):
  • Study Protocol (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT03879668/Prot_000.pdf